CLINICAL TRIAL: NCT01274195
Title: Hematopoietic Stem Cell Transplantation With Targeted Busulfan and Fludarabine in Pediatric AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUCH-SCT -1001
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic stem cell transplantation
MeSH Terms: interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Busulfan (Experimental)
  Interventions: Drug: Busulfan

INTERVENTIONS:
Drug: Busulfan — First dose: busulfan (120 mg/m2 ivs once daily) (if age<1 yr: 80 mg/ m2) Second to forth dose: according to the daily pharmacokinetic study

SUMMARY:
In this study we plan to improve the outcome of hematopoietic stem cell transplantation by using optimal busulfan dose through pharmacokinetic study.

DETAILED DESCRIPTION:
Busulfan is a highly toxic drug with narrow therapeutic window used for the conditioning of hematopoietic stem cell transplantation. High exposure is associated with systemic toxicity such as veno-occlusive disease (VOD) and underexposure is associated with graft failure or relapse. In this study the investigators plan to improve the outcome of hematopoietic stem cell transplantation by using optimal busulfan dose through pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed as AML.
2. Patients who need hematopoietic stem cell transplantation with busulfan based conditioning regimen.
3. Age: up to 21 years
4. Performance status: ECOG 0-2.
5. Patients must be free of significant functional deficits in major organs, but the following eligibility criteria may be modified in individual cases. 1. Heart: a shortening fraction > 30% and ejection fraction > 45%. 2. Liver: total bilirubin < 2 × upper limit of normal; ALT < 3 × upper limit of normal. 3. Kidney: creatinine <2 × normal or a creatinine clearance (GFR) > 60 ml/min/1.73m2.
6. Patients must lack any active viral infections or active fungal infection.
7. Appropriate donor is available: Matched in 6/6 of A, B, DR loci.
8. Patients (or one of parents if patients age < 20) should sign informed consent.

Exclusion Criteria:

1. Pregnant or nursing women.
2. Malignant or nonmalignant illness that is uncontrolled or whose control may be jeopardized by complications of study therapy.
3. Psychiatric disorder that would preclude compliance.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate 1-year event free survival after hematopoietic stem cell transplantation. | For 4 days used Buslufan through pharmacokinetic study in hematopoietic stem cell transplantation
  To evaluate 1-year event free survival after hematopoietic stem cell transplantation.

SECONDARY OUTCOMES:
To evaluate engraftment rate, toxicities associated with hematopoietic stem cell transplantation, acute and chronic GVHD, treatment related mortality and relapse rate. | 1, 3, 6 and 12 months after transplantation
  To evaluate engraftment rate, toxicities associated with hematopoietic stem cell transplantation, acute and chronic GVHD, treatment related mortality and relapse rate.

CONTACTS AND LOCATIONS:
Overall Officials: Hyoung Jin Kang, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Daehangno, Jongno-gu, South Korea